CLINICAL TRIAL: NCT04827368
Title: Non-invasive Disease Activity Monitoring in Patients With Inflammatory Bowel Disease (IBD) Using Volatile Organic Compounds
Brief Title: Volatile Organic Compounds (VOCs) in Active Inflammatory Bowel Disease
Acronym: VOC
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Florian Rieder, Principal Investigator, The Cleveland Clinic
Other Study IDs: 20-1149; B19-566 (Other: Abbvie)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: IBD; Crohn Disease; Ulcerative Colitis
Keywords: IBD, VOC
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum: Will be obtained from whole blood Stool: will be collected using standard collection containers and procedures and aliquoted Breath: Subjects will be nil per orally (NPO) for 8 hours prior to breath collection and they will rinse their mouths and gargle with water immediately before obtaining the breath sample to eliminate contamination from oral VOCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Crohns Disease: Potential participants will be identified based on their planned/scheduled endoscopy visit.
  Interventions: Other: Breath Test
- Ulcerative Colitis: Potential participants will be identified based on their planned/scheduled endoscopy visit.
  Interventions: Other: Breath Test
- Non-IBD: Healthy subjects with no bowel disorders will be included as controls.
  Interventions: Other: Breath Test

INTERVENTIONS:
Other: Breath Test — Research Breath sample through disposable mouth filter. Serum sample through routine blood draw. Stool sample through standard collection containers.
  Other Names: Serum Samples; Stool Samples

SUMMARY:
Inflammatory Bowel Disease (IBD) are chronic diseases of the gut comprising Crohn's Disease (CD) and Ulcerative Colitis (UC). The symptoms of IBD consist of diarrhea, abdominal discomfort, weight loss, fatigue and rectal bleeding. However, symptoms and treatment vary between patients. Early management of IBD can lead to better response rates and decrease the risk of irreversible bowel damage and future disease complications such as surgeries. Current clinical tools for diagnosis and or assessing progression of IBD are either invasive (colonoscopy), have low patient acceptance (fecal calprotectin) or low accuracy (C-reactive protein). The purpose of this study is to collect clinical data and samples (including blood, breath and stool) donated by patients with IBD and patients with no IBD (controls) to facilitate research that may result in the development of new non-invasive methods of diagnosing IBD and understand the progression of the disease over time in order to better manage IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having Crohn's Disease or Ulcerative Colitis
* Aged 18-70 years.
* Understands the language and signs an informed consent form.
* Any disease location, except isolated upper GI Crohn's disease only
* Any CD or UC disease activity.
* Outpatients and inpatients
* Patients will be recruited, and samples obtained at least one day, and no more than one week, prior to out/inpatient colonoscopy preparation to allow objective assessment of disease activity.

Exclusion Criteria:

* Status post colectomy
* Status post diverting loop ileostomy or end ileostomy or colostomy
* On antibiotics in the past 3 months or currently
* Women (pregnant or breast feeding)
* Subjects with concurrent chronic liver, renal, lung or metabolic disorders
* Active malignancy
* Bowel preparation at day of sample procurement
* Isolated upper GI Crohn's disease only
* Active disease on colonoscopy, but normal fecal calprotectin at inclusion
* C diff. positive at time of inclusion (test to be obtained in routine clinical care).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, controlled, non-interventional cohort study, conducted at the Cleveland Clinic IBD Center, using serially obtained breath and serum headspace VOCs as non-invasive biomarkers to detect disease activity in IBD, fecal calprotectin, CRP, and patient-reported outcome tools. No drug will be evaluated in this study. All visits for this study as well as the initial endoscopy will be based on standard clinical practice and guidelines.
  At inclusion, all patients will have a colonoscopy (indication is standard of care), CRP, fecal calprotectin, and baseline PRO2 to establish the pattern for disease activity, which will subsequently be evaluated for change by using fecal calprotectin, CRP, and PRO2 over one year (every 3 months), as a surrogate marker for disease activity.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Breath volatile organic compounds (VOC)s and objective markers of Inflammatory Bowel Disease (IBD) Activity | 1 year
  Correlation of breath VOCs with changes in Fecal Calprotectin.

SECONDARY OUTCOMES:
Breath volatile organic compounds (VOC)s and objective markers of Inflammatory Bowel Disease (IBD) Activity | 1 year
  Correlation of breath VOCs with changes in C-reactive protein (CRP) and clinical disease activity

OTHER OUTCOMES:
Breath volatile organic compounds (VOC)s and objective markers of Inflammatory Bowel Disease (IBD) Activity | 1 year
  Correlation of breath VOCs with endoscopic disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Florian Rieder, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States